CLINICAL TRIAL: NCT00080093
Title: Increasing Condom Use With a Stage-Matched Intervention
Brief Title: Increasing Condom Use in People at Risk for HIV Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Patricia Morokoff, PhD, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AI041323 (NIH); R01AI041323 (NIH)
Record Dates: First submitted 2004-03-23; First posted 2004-03-24 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Condom; HIV Seronegativity; HIV Prevention; Behavioral Intervention
MeSH Terms: conditions — HIV Infections

ARMS (2):
- 1 (Experimental): Participants will receive individual feedback and specially-tailored manuals at study entry and at Months 2 and 4
  Interventions: Behavioral: Individual feedback and specially-tailored manuals
- 2 (Experimental): Participants will receive general HIV information feedback and the best-available informational manual at study entry and at Months 2 and 4
  Interventions: Behavioral: General HIV information feedback and the best-available information

INTERVENTIONS:
Behavioral: Individual feedback and specially-tailored manuals — Individual feedback and specially-tailored manuals
  Arms: 1
Behavioral: General HIV information feedback and the best-available information — General HIV information feedback and the best-available information
  Arms: 2

SUMMARY:
This study will evaluate a new program designed to increase condom use in both women and men.

DETAILED DESCRIPTION:
As heterosexual HIV transmission increases, effective behavioral interventions to increase condom use are needed. Interventions should be low cost and accessible to large segments of the at-risk population. This study will evaluate the efficacy of a behavioral intervention designed to increase condom use in at-risk, heterosexually active women and men. The intervention is computer-delivered and will be provided in health care settings. The study will also examine additional psychosocial mediators of condom use by testing the predictive efficacy of the Multifaceted Model of HIV Risk.

Participants will be recruited from four health clinic sites that serve local ethnic minority communities. The participants will be randomly assigned to either an individualized intervention designed to increase condom use or to an HIV information comparison group. All participants will receive comparable group-specific informational materials at study entry and at Months 2 and 4. Participants in the intervention group will receive individualized feedback and specially-tailored manuals. Participants in the HIV information comparison group will receive general HIV information feedback and the best-available informational manual.

Assessments for both groups will be conducted at study entry and at Months 6, 12, and 18. At study entry, participants will complete paper and pencil questionnaires lasting about 30 minutes. There will also be computer question sessions at study entry and at Months 2 and 4. Participants will be asked about condom use, contraceptive use, risk behaviors, sexual transmitted disease (STD) history, and personal relationships. Telephone follow-ups at Months 6, 12, and 18 will take approximately 20 to 30 minutes.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected
* Sexually active
* At risk for HIV (as determined by study officials)
* Speaks English
* Seen at a participating clinic

Exclusion Criteria

* Pregnant

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 534 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of condom use | At 30 days and 2 months before each assessment
Number of occurances of unprotected sex | At 30 days before each assessment
Stage of change for condom use with main and nonmain partners, and men and women | Throughout study

SECONDARY OUTCOMES:
Frequency of condom use with main and nonmain partners, and men and women | Throughout Study
Number and ratios of protected sex occasions with main and nonmain partners, and men and women | Throughout study
Stage of change for condom use with main and nonmain partners, and men and women | Throughout Study

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Morokoff, PhD, Principal Investigator — University of Rhode Island

REFERENCES:
- [Result] Cho S, Harlow L, Morokoff P, Redding C, Rossi J, Mayer K, Koblin B. Predicting 3-Wave LGCM of Condom Use in High-Risk Community Sample. Annual Meeting of the American Psychological Association, San Francisco, CA, 2007.
- [Result] Cho S, Morokoff P, Redding C, Harlow L, Rossi J, Mayer K, Koblin B. Empirically Investigating Gender in a Multifaceted Model of HIV Risk. 19th Annual Meeting of the American Psychological Society, Washington, DC, 2007.